CLINICAL TRIAL: NCT01368094
Title: Early (4 Days) Versus Standard Drainage Removal of the Abdominal Cavity After Pancreaticoduodenectomy- - A Randomized Multicenter Study
Brief Title: Early (4 Days) Versus Standard Drainage of the Abdominal Cavity After Pancreaticoduodenectomy
Acronym: DRAINAGE DPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRCIR10-PR-REGIMBEAU; 2010-A01347-32 (Other: ID-RCB)
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Disease; Pancreatic Neoplasms
Keywords: Pancreaticoduodenectomy; Drainage; Surgical site infection
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard drainage (Active Comparator)
  Interventions: Procedure: Standard drain removal
- Short drainage (Experimental)
  Interventions: Procedure: Drain removal at D4

INTERVENTIONS:
Procedure: Drain removal at D4 — If no pancreatic fistula (PF) or deep SSI is highlighted neither on the CT-scanner nor with biological analysis, on day 3 postoperatively, the drain will be removed on the 4th postoperative day, at the patient's bedside.
  Arms: Short drainage
Procedure: Standard drain removal — If no pancreatic fistula (PF) or deep SSI is highlighted on the CT-scanner on day 3 postoperatively, the drain will be removed following the clinical routine practice of the surgical team that takes the patient in charge. The patient will leave the department when the surgeon deems necessary.
  Arms: Standard drainage

SUMMARY:
Around two thousand pancreaticoduodenectomy (PD) are performed each year in France. This intervention is associated with a high rate of postoperative complications including:

* pancreatic fistulas (PF);
* surgical site infections (intra-abdominal abscess, wound infection);
* delayed gastric emptying (gastroparesis);
* and hemorrhage.

The incidence of SSI (superficial and deep) is about 35% and seems influenced by the prolonged intra-abdominal drainage. For several years, there has been a global trend to reduce the use of abdominal drainage after abdominal surgery. Several randomized clinical trials have shown that prophylactic drainage does not decrease the incidence of postoperative complications during elective hepatectomy, colectomy, and cholecystectomy and could increase the number of SSI. However, the role of prophylactic drainage after PD is so far unclear.

The aim of this prospective randomized multicenter study is to evaluate the influence of early (4 days) versus standard (10 to 15 days, depending on the staff clinical practice) drainage removal of the abdominal cavity after PD, on the rate of SSI.

Materials and Methods: The technique of PD is left at the discretion of the operator as well as the prescription of analogues of somatostatin. Drainage of the abdominal cavity is made of one or two round silicone close suction drains or open multichannel silicone drains placed in the vicinity of the pancreatic and biliary anastomosis. Shall be excluded patients operated on for chronic pancreatitis and patients who underwent preoperative radiotherapy. The 3rd postoperative day, a fistula is sought clinically, biologically and on CT-scanner images. In case of pancreatic fistula, the patient is excluded from randomization and drainage of the abdominal cavity is left in place depending on the different teams' practice. Patients without fistula are randomized to either drainage removal 4 days after surgery (D4) or standard drainage.

DETAILED DESCRIPTION:
Introduction. Two thousand pancreaticoduodenectomy (PD) are performed per year in France (observatory pancreatectomy GCB 2005). This intervention is associated with a high rate of postoperative complications including pancreatic fistula (PF), the site infections (SSI: intra-abdominal abscess, wound infection), gastroparesis, and hemorrhage. The incidence of SSI (superficial and deep) is about 35% and seems influenced by the prolonged drainage of intra-abdominal. For several years, there is a global trend to reduce the use of abdominal drainage after abdominal surgery. Several randomized clinical trials have shown that prophylactic drainage does not decrease the incidence of postoperative complications during elective hepatectomy, colectomy, and cholecystectomy and could increase the number of SSI. However, the role of prophylactic drainage after PD is so far unclear. In the literature, three studies have examined the influence of drainage of the abdominal cavity after PD, and were published at the time this protocol was submitted :

* The study of Conlon et al. (Ann Surg 2001), prospective randomized study comparing no drainage standard abdominal drainage. The SSI rates in the drained group was 36% versus 16% in the undrained group (NS, but in his critical study methodology).
* The study of Kawai et al. (Ann Surg 2006), non-randomized prospective study comparing short drainage (D4) drainage standard (D8). The SSI rates in the drained group was 38% versus 7.7% in the undrained group (significant but non-randomized study involving patients on two consecutive periods).
* Study Berberat et al. (Büchler) (J Gastrointest Surg 2007), retrospective analysis of a population of patients with a PD (80%) the results by intention to treat the early removal of drainage of the abdominal cavity. The SSI rates published in this study is 9.4%.

After acceptance of this protocol by local ethics committee, a forth study was published by Bassi et al (Bassi C Ann Surg 2010) : it is a randomized controlled study. Patients who underwent pancreatic resection (including left pancreatic resection) and at low risk of postoperative pancreatic fistula were randomized on post operative day (POD) 3 to receive either early (POD 3) or standard drain removal (POD 5 or beyond). The primary end point of the study was the incidence of pancreatic fistula. This study shows that, in patients with a low risk of pancreatic fistula after pancreatic resection, intra-abdominal drains can be safely removed on POD 3 after standard pancreatic resections. A prolonged period of drain insertion is associated with a higher rate of postoperative complications with increased hospital stay.

The aim of the present prospective randomized multicenter study is to evaluate the influence of short drainage (4 days) of the abdominal cavity versus standard drainage (10 to 15 days, depending on the staff clinical practice) after PD on the rate of SSI.

Materials and Methods: The technique of PD is left at the discretion of the operator as well as the prescription of analogues of somatostatin. Drainage of the abdominal cavity is made of one or two round silicone close suction drains or open multichannel silicone drains placed in the vicinity of the pancreatic and biliary anastomosis. Shall be excluded patients operated on for chronic pancreatitis and patients who underwent preoperative radiotherapy. The 3rd postoperative day, a pancreatic fistula is sought clinically, biologically and on CT-scanner images. In case of pancreatic fistula, the patient is excluded from randomization and drainage of the abdominal cavity is left in place depending on the different teams' practice. Patients without fistula are randomized to either drainage removal 4 days after surgery (D4) or standard drainage.

Analysis and outcomes: The primary endpoint will be the occurrence of surgical site infection (SSI) at D30, as defined by:

* surface SSI (wound abscess): infection of the skin, subcutaneous tissue or muscle, above the fascia, located at a surgical incision. The diagnosis is based on at least one of the following criteria:

  * The fluid from the wound or drain located above the fascia is purulent
  * A spontaneous dehiscence of the wound
  * A positive culture from a closed wound.
* deep SSI (intra-abdominal abscess) infection in operated tissues or in site of intervention (under the fascia). The diagnosis is based on at least one of the following criteria:

  * The fluid from a drain positioned beneath the fascia is purulent;
  * A culture from a closed wound is positive;
  * Other signs of infection on direct examination found during a re-operation.

Secondary outcomes will be the length of hospital stay, postoperative complications, with emphasis on classification IIIa (radiological drainage) and IIIb (re-intervention) of Clavien (Dindo et al. Ann Surg 2004).

All patients who underwent PD during the study period, especially patients excluded before randomization will be collected.

Calculating the number of patients needed to reduce SSI rate from 30% (in the group standard drainage of the abdominal cavity) to 10% (in the short drainage group), with a risk alpha of 0.05 and a risk beta of 0.20 yields 124 patients. Taking into account 10% of patients not analyzable, the number of patients included in this study is 138 (69 patients in each arm).

Five university hospitals are participating in the study (Amiens, Lille, Caen, and Rouen) and one general hospital (CH Beauvais). The expected duration of the study is 24 months (12-14 patients per center per year).

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic tumor regardless of its nature: All patients requiring PD (following thesaurus or multidisciplinary team council recommendation) for this indication will be included.
* Ability to participate in a clinical research protocol.
* Given informed consent.

Exclusion Criteria:

* History of pancreatic surgery or biliary diversion and / or digestive
* Patient taken in charge for chronic pancreatitis without tumor
* History of supramesocolic radiotherapy
* Sick supported emergency
* Physical or mental condition does not allow participation in the study
* Contra-indication to surgery
* ASA classification (American Society of Anesthesiologists) IV-V or life expectancy <48
* Pregnancy or breastfeeding
* Patient under guardianship or private patient of liberty by a judicial or administrative decision
* Age under 18yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection at D30 | 30 days after surgical intervention
  The outcome measure is the occurrence of surgical site infection (SSI) at D30, as defined by:
  * surface SSI (wound abscess): infection of the skin, subcutaneous tissue or muscle, above the fascia, located at a surgical incision.
  * deep SSI (intra-abdominal abscess) infection in operated tissues or in site of intervention (under the fascia).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc REGIMBEAU, Pr, Principal Investigator — Centre Hospitalier Régional Universitaire d'Amiens
Locations (5):
- France (5):
  - CHU Amiens, Amiens, Picardie
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier Saint-Martin, Caen
  - Centre Hospitalier Régional Universitaire Claude Huriez, Lille
  - Centre Hospitalier Charles Nicolle, Rouen

REFERENCES:
- [Result] Dembinski J, Mariette C, Tuech JJ, Mauvais F, Piessen G, Fuks D, Schwarz L, Truant S, Cosse C, Pruvot FR, Regimbeau JM. Early removal of intraperitoneal drainage after pancreatoduodenectomy in patients without postoperative fistula at POD3: Results of a randomized clinical trial. J Visc Surg. 2019 Apr;156(2):103-112. doi: 10.1016/j.jviscsurg.2018.06.006. Epub 2019 Jan 31. PMID 30713100